CLINICAL TRIAL: NCT00659373
Title: Investigating Cognitive Function for Patients Participating in the SOFT Trial in Selected Centers
Brief Title: Brain Function in Premenopausal Women Receiving Tamoxifen With or Without Ovarian Function Suppression for Early-Stage Breast Cancer on Clinical Trial IBCSG 24-02
Acronym: Co-SOFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Breast Cancer Trials, Australia and New Zealand (Other); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CDR0000594003; IBCSG-24-02-ANZ0701; ANZ0701; CALGB-IBCSG-24-02-ANZ0701
Record Dates: First submitted 2008-04-15; First posted 2008-04-16 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Fatigue; Sleep Disorders
Keywords: cognitive/functional effects; psychosocial effects of cancer and its treatment; fatigue; sleep disorders; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Sleep Wake Disorders | interventions — Tamoxifen; Triptorelin Pamoate; Gonadotropin-Releasing Hormone; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tamoxifen (Active Comparator): Tamoxifen 20mg orally daily for 5 years
  Interventions: Drug: Tamoxifen
- T+OFS (Experimental): Tamoxifen 20mg orally daily for 5 years plus ovarian function suppression (OFS; triptorelin (GnRH analogue) 3.75 mg by im injection q28 days for 5 years; or surgical oophorectomy; or ovarian irradiation)
  Interventions: Drug: Tamoxifen; Drug: triptorelin
- E+OFS (Experimental): Exemestane 25mg orally daily for 5 years plus ovarian function suppression (OFS; triptorelin (GnRH analogue) 3.75 mg by im injection q28 days for 5 years; or surgical oophorectomy; or ovarian irradiation)
  Interventions: Drug: triptorelin; Drug: Exemestane

INTERVENTIONS:
Drug: Tamoxifen
  Other Names: Nolvadex
  Arms: T+OFS; Tamoxifen
Drug: triptorelin
  Other Names: GnRH analogue; Trelstar Depot; Decapeptyl Depot
  Arms: E+OFS; T+OFS
Drug: Exemestane
  Other Names: Aromasin
  Arms: E+OFS

SUMMARY:
RATIONALE: Learning about the long-term effects of adjuvant tamoxifen (T), adjuvant tamoxifen with ovarian function suppression (T+OFS), and exemestane with ovarian function suppression (E+ OFS) on brain function may help doctors plan cancer treatment.

PURPOSE: This study is looking at brain function in premenopausal women who are receiving adjuvant tamoxifen (T) alone against those receive adjuvant tamoxifen (T+OFS) or exemestane (E+OFS) with ovarian function suppression (OFS) for early-stage breast cancer on clinical trial IBCSG-2402.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

* To evaluate and compare the changes in cognitive function over one year in premenopausal breast cancer patients who receive adjuvant tamoxifen (T) alone against those receive adjuvant tamoxifen (T+OFS) or exemestane (E+OFS) with ovarian function suppression (OFS).

OUTLINE: This is a multicenter study.

Objective cognitive function was measured with the CogState computerized test battery. The CogState battery consists of seven tasks: Detection, Identification, Monitoring, Memory, Learning, International Shopping List Task (ISLT), and ISLT-Delayed Recall. Performance speed is measured for the Detection, Identification and Monitoring tasks and performance accuracy is measured for the Memory, Learning, ISLT, and ISLT-Delayed Recall. Measures of performance speed are normalized using measures of performance accuracy (%) are normalized using arcsine transformation. The main outcome measure is a composite score which is the average of these task scores (after transformation and standardization by age-specific norms). Patients complete these assessments at baseline (i.e. before start of protocol hormonal therapy) and approximately one year after randomization to the parent IBCSG 24-02 (SOFT) study.

Data were collected separately for the T+OFS and E+OFS participants in the parent study, IBCSG 24-02 (SOFT). The sample size for this Co-SOFT substudy was small, so the analysis plan was revised to pre-specify collective analysis for all patients receiving OFS.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Completely resected disease
* Registered for clinical trial IBCSG-2402, but not yet started protocol hormonal therapy

  * Has not yet received any of the following adjuvant endocrine therapy, either before or after registration on IBCSG-2402:

    * Tamoxifen, exemestane, or gonadotropin-releasing hormone (GnRH) agonist
    * Ovarian irradiation
    * Bilateral oophorectomy
* Hormone receptor status:

  * Estrogen and/or progesterone receptor positive

    * Each tumor must be hormone receptor positive

PATIENT CHARACTERISTICS:

* Premenopausal
* Can speak and read the local language(s) fluently

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-12; Primary Completion 2014-12 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juerg Bernhard, PhD, Study Chair — ETOP IBCSG Partners Foundation; Kelly-Anne Phillips, Study Chair — Peter MacCallum Cancer Centre, Australia; Timothy Ahles, MD, Study Chair — Cancer and Leukemia Group B
Locations (15):
- United States (13):
  - Mercy General Hospital, Sacramento, California
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
- Canada (2):
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario

REFERENCES:
- [Result] Phillips KA, Regan MM, Ribi K, Francis PA, Puglisi F, Bellet M, Spazzapan S, Karlsson P, Budman DR, Zaman K, Abdi EA, Domchek SM, Feng Y, Price KN, Coates AS, Gelber RD, Maruff P, Boyle F, Forbes JF, Ahles T, Fleming GF, Bernhard J. Adjuvant ovarian function suppression and cognitive function in women with breast cancer. Br J Cancer. 2016 Apr 26;114(9):956-64. doi: 10.1038/bjc.2016.71. Epub 2016 Apr 19. PMID 27092785

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data were collected separately for the T+OFS and E+OFS participants in the parent study, IBCSG 24-02 (SOFT). The sample size for this Co-SOFT substudy was small, so the analysis plan was revised to pre-specify collective analysis for all patients receiving OFS.
Groups:
- Ovarian Function Suppression: Tamoxifen 20mg orally daily or Exemestane 25mg orally daily for 5 years plus ovarian function suppression (OFS; triptorelin (GnRH analogue) 3.75 mg by im injection q28 days for 5 years; or surgical oophorectomy; or ovarian irradiation)
Period: Overall Study
Arm/Group | Tamoxifen | Ovarian Function Suppression
Started | 25 | 61
Completed | 20 | 54
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Assessment Missed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Ovarian Function Suppression: Tamoxifen 20mg orally daily or Exemestane 25mg orally daily for 5 years plus ovarian function suppression (OFS; triptorelin (GnRH analogue) 3.75 mg by im injection q28 days for 5 years; or surgical oophorectomy; or ovarian irradiation).
  Note: Data were collected separately for the T+OFS and E+OFS participants in the parent study, IBCSG 24-02 (SOFT). The sample size for this Co-SOFT substudy was small, so the analysis plan was revised to pre-specify collective analysis for all patients receiving OFS.
- Total: Total of all reporting groups
Arm/Group | Tamoxifen | Ovarian Function Suppression | Total
Number analyzed (Participants) | 20 | 54 | 74
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [43 to 50] | 45 [41 to 47] | 45 [41 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 54 | 74
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function Over 1 Year in Premenopausal Breast Cancer Patients Who Receive Adjuvant Tamoxifen (T) Alone Against Those Receive Adjuvant Tamoxifen (T+OFS) or Exemestane (E+OFS) With Ovarian Function Suppression (OFS)
Description: Objective cognitive function measured with CogState, a computerized test battery of 7 tasks: Detection, Identification, Monitoring, Memory, Learning, International Shopping List Task (ISLT) and ISLT-Delayed Recall. Performance speed is measured for Detection/Identification/Monitoring and performance accuracy is measured for Memory/Learning/ISLT/ISLT-Delayed Recall. Performance speed calculated as mean of the log10 transformed reaction time for correct responses (lower score=better); performance accuracy calculated as arcsine transformation of the proportion of correct responses (higher scores=better). Main outcome measure is a composite score (average of task scores after transformation and standardization by age-specific norms). A positive standardized score indicates that a patient performed better than average; a negative standardized score indicates below average results. Patients complete assessments at baseline and 1 year after randomization to parent IBCSG 24-02 (SOFT) study.
Time Frame: 1 year after patient randomization to parent IBCSG 24-02 study
Measure: Mean (Standard Deviation); unit: standardized units
Groups:
- Ovarian Function Suppression: Tamoxifen 20mg orally daily or Exemestane 25mg orally daily for 5 years plus ovarian function suppression (OFS; triptorelin (GnRH analogue) 3.75 mg by im injection q28 days for 5 years; or surgical oophorectomy; or ovarian irradiation)
  Note: Data were collected separately for the T+OFS and E+OFS participants in the parent study, IBCSG 24-02 (SOFT). The sample size for this Co-SOFT substudy was small, so the analysis plan was revised to pre-specify collective analysis for all patients receiving OFS.
Arm/Group | Tamoxifen | Ovarian Function Suppression
Number analyzed (Participants) | 20 | 54
standardized units | -.04 (0.49) | -0.21 (0.92)
Statistical Analysis 1: Comparison: Tamoxifen vs Ovarian Function Suppression; Test type: Superiority or Other; p = 0.71, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Tamoxifen | Ovarian Function Suppression
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/54
Other Adverse Events (participants affected / at risk) | 0/20 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No